CLINICAL TRIAL: NCT05469490
Title: Phase I Study Investigating the Safety of Navoximod and NLG802 in Combination With Stereotactic Body Radiotherapy (SBRT) in Subjects With Advanced Solid Tumors
Brief Title: Safety of Navoximod and NLG802 With Stereotactic Body Radiotherapy (SBRT) Treatment of Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding support.
Sponsor: Luke, Jason, MD (Other)
Collaborators: Lumos Pharma (Industry)
Responsible Party: Principal Investigator, Adam Olson, Clinical Assistant Professor of Medicine, Department of Radiation Oncology, UPMC Hillman Cancer Center, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-257
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumors
Keywords: Stereotactic Body Radiotherapy (SBRT); immune-oncology (IO) agents; Indoleamine 2,3-dioxygenase 1 (IDO1)
MeSH Terms: interventions — Radiosurgery; navoximod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) + NLG802 and navoximod (Experimental): SBRT - Initial Starting Dose:
  Lung - Peripheral - 45 Gy (3 fractions) Lung - Central OR Mediastinal/Thoracic/Axillary/Cervical Lymph Node - 50 Gy (5 fractions) Liver - 45 Gy (3 fractions) Spinal/Paraspinal OR Osseous - 30 Gy (3 fractions) Abdominal/Pelvic (including Adrenal Gland) - 45 Gy (3 fractions)
  SBRT - Decreased DLT Dose:
  Lung - Peripheral - 42 Gy (3 fractions) Lung - Central OR Mediastinal/Thoracic/Axillary/Cervical Lymph Node - 47.5 Gy (5 fractions) Liver - 42 Gy (3 fractions) Spinal/Paraspinal OR Osseous - 27 Gy (3 fractions) Abdominal/Pelvic (including Adrenal Gland) - 42 Gy (3 fractions)
  NLG802 - 1452mg BID (no dose decrease)
  navoximod - Starting dose: 1000mg BID, Dose decrease 1: 800mg BID, Dose decrease 2: 600mg BID
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT); Drug: navoximod; Drug: NLG802 (indoximod Prodrug)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT is specialize radiation that is effective for ablating tumors at primary and metastatic locations that increases antigen uptake/processing/presentation.
Drug: navoximod — A small molecule inhibitor with potent inhibition of IDO1 enzymatic activity as shown both in vitro and in vivo. As the main function of IDO1 is the regulation of acquired immune tolerance, and its expression in tumor- and dendritic cells in tumor draining lymph nodes negatively correlates with cancer prognosis and survival, navoximod-mediated IDO1 inhibition may restore immune reactivity towards tumors.
  Other Names: (GDC-0919; previously NLG919)
Drug: NLG802 (indoximod Prodrug) — An anti-tumor immunomodulator with the active ingredient of 1-methyl-D-tryptophan (NSC- 721782, 1-MT), which is an inhibitor of the indoleamine 2,3-dioxygenase (IDO) pathway that increases the bioavailability of indoximod by leveraging existing mechanisms of absorption, increasing the exposure of indoximod.

SUMMARY:
This early phase trial proposes to study of stereotactic body radiation therapy (SBRT) with navoximod and NLG802, a prodrug of indoximod. Combinations of immune-oncology (IO) agents with complementary mechanisms as well as radiation represent a promising strategy to improve response rates to immunotherapy. Radiation therapy induces immunogenic cell death, increases production of tumor specific antigens, enhances TH cell functioning, and modulates immunosuppressive cell populations such as T regulatory cells and myeloid derived suppressor cells.

DETAILED DESCRIPTION:
Treatment for this trial will include stereotactic body radiation therapy (SBRT) to 1-4 metastases that can be safely irradiated, in combination with NLG802 and navoximod. The study will determine the safe doses of SBRT in combination with navoximod and NLG802 twice per day. The amount of SBRT administered will range from 30Gy to 50 Gy, depending upon the location of the tumor. If dose-limiting toxicities (DLT) are experienced, SBRT will be decreased accordingly. Disease assessment with computed tomography (CT) and/or magnetic resonance imaging (MRI if CT scan is contraindicated) will be performed in the screening period, after 8 weeks of starting SBRT/NLG802/navoximod and then every 8 weeks until progression of disease, at the completion of follow-up, or until participants withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor for which curative treatment is not available
* Undergone appropriate standard of care treatment options (in the opinion of the treating investigator).
* Evaluable disease by serum tumor marker or measurable disease as defined by RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Adequate organ function, as defined by the following:

  * Absolute neutrophil count (ANC) ≥ 1,500/μL
  * Platelets ≥ 100×10^3/μL
  * Hemoglobin ≥ 8 g/dL
  * Serum creatinine ≤ 1.5× institutional upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCL) > 50 mL/min (creatinine clearance should be calculated per institutional standard). GFR can also be used in place of creatinine of CrCl.
  * Serum total bilirubin ≤1.5× institutional ULN (except subjects with Gilbert's Syndrome, who must have normal direct bilirubin).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× institutional ULN OR < 5x ULN for subjects with liver metastases.
  * Albumin > 3.2 mg/dL.
* Participants may have had prior IO therapy (including but not limited to anti-CTLA4 and anti-PD1/L1) excluding prior IDO inhibitors

Age and Reproductive Status

* Males and females ≥ 15 years of age at the time of informed consent.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) or serial HCG at least one week apart demonstrating no rise consistent with pregnancy prior to the start of study drug.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 5 months post last dose of study drug(s).
* WOCBP who are continuously not heterosexually active are exempted from contraceptive requirements but still must undergo pregnancy testing as described in this section.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 7 months post last dose of study drug(s).
* Male participants must be willing to refrain from sperm donation during this time.
* Azoospermic males are exempt from contraceptive requirements. Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy.

Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly.

Exclusion Criteria:

* Currently receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 or have not recovered (i.e. < grade 1 at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, radiation or other anti-cancer therapy (with exceptions for disease-specific hormone treatments considered standard of care) within 2 weeks prior to study Day 1 or have not recovered (i.e. < grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: subjects with < grade 2 neuropathy, endocrinopathy which is adequately controlled with hormone replacement therapy are an exception to this criterion and may qualify for the study.
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Symptomatic or clinically relevant active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Patients with asymptomatic brain lesions deemed clinically irrelevant by the treating investigator are allowed.
* Prior radiation therapy (defined as >10% of prior prescription dose) to the area planning to be treated with radiation.
* Diagnosis of immunodeficiency or are receiving systemic steroid therapy at a dose of >10 mg prednisone daily or equivalent at time of first dose of trial treatment for another reason.
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity or history of allergy to NLG802 and navoximod
* Known additional malignancy that could confuse analysis of on-study treatment. Inclusion of all study participants with more than one malignancy must be discussed and approved by the PI.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of non-infectious pneumonitis that required steroids for treatment.
* Evidence of interstitial lung disease.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known active psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) then patient is not eligible for cohorts including SBRT to liver lesions.
* Prior organ allograft or allogeneic bone marrow transplantation.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke with clinical sequalae within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes). Controlled atrial fibrillation is allowed.
  * History of other clinically significant heart disease (e.g., cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
* Received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. COVID-19 vaccination is allowed.
* Participants must not be prisoners or be involuntarily incarcerated.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 90 days (patient)
  The RP2D is determined by the occurrence of Dose-limiting Toxicities (DLT) defined as any Grade 3 or 4 toxicities to relevant organ systems determined to be possibly, likely or definitely related to treatment, deemed by the treating investigator that further administration of NLG802 and navoximod as not considered to be safe. Grade 3: Hold both NLG802 and navoximod until the AE recovers to Grade 0-1 or to pretreatment baseline level, whichever is more severe, and then resume treatment with NLG802 and navoximod at a dose level reduction. Clinically insignificant grade 3 events (ie - amylase/lipase) do not require drug hold Grade 4: Discontinue all study treatment permanently and withdraw patient from the study. Toxicity will be attributed to the combination of radiation with immunotherapy (as opposed to individual elements).If a dose reduction is required because of treatment-related toxicities, no dose re-escalation will be permitted for the duration of study treatment.

SECONDARY OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 1 year (patient), up to 4 years (cohort)
  The number of patients incurring specific Adverse Events or Serious Adverse Events that occur from first day of treatment, considered to be possibly, probably or definitely related to study treatment, per Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Patients experiencing multiple AEs of the same type will be reported by only the most severe grade.
Objective response rate (ORR) | Up to 1 year (patient), up to 4 years (cohort)
  The proportion of patients with complete or partial response per iRECIST. irCR (Complete Response):Disappearance of non-nodal lesions. All pathologic lymph nodes <10 mm (2 consecutive measures ≥4 weeks apart); irPR (Partial Response):≥30% decrease from baseline (2 consecutive measures ≥4 weeks apart); All pathologic lymph nodes <10 mm (Non-Target Lesions: Any other than disappearance of all non-nodal lesions and reduction of pathologic lymph nodes <10 mm). Baseline tumor burden: sum of single diameters (short axis for nodal lesions, longest diameter for other lesions) for target lesions. In subsequent scans, the diameters of new measurable lesions are added to the tumor burden. Re-treatment: ≤5 target lesions (=/≠ original lesions) are selected and a new baseline tumor burden will be established.
Progression-free survival (PFS) | Up to 4 years
  The number of months from the date of study enrollment to the date of an event of disease progression (per RECIST 1.1) or to the date of death from any cause. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Up to 4 years
  The number of months from the date of study enrollment until date of death ( from any cause) or last known date of follow up if otherwise lost to follow up.
Local control per RECIST version 1.1 | Up to 4 years
  Proportion of patients without disease progression in area of RT treatment. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Local control by irRECIST | Up to 4 years
  Proportion of patients without disease progession in the area of RT treatment. Progressive Disease (iCPD) per iRECIST is present if further progress of the target sum (≥ 5 mm), or any further progress of the Non-Target Lesion, and/or progress of the new measurable and not measurable lesions either in number or in size (sum ≥5 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Olson, MD, MS, Principal Investigator — UPMC Hillman Cancer Center

IPD SHARING:
Plan to Share IPD: No